CLINICAL TRIAL: NCT00448214
Title: Direct Factor Xa Inhibitor YM150 for Prevention of Stroke in Subjects With Non-Valvular Atrial Fibrillation - A Double Blind, Parallel, Dose-finding Study in Comparison With Open Label Warfarin
Brief Title: Direct Factor Xa Inhibitor YM150 for Prevention of Stroke in Subjects With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 150-CL-030
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Atrial Fibrillation
Keywords: Factor Xa inhibitor; Atrial fibrillation; Stroke; Ischemic attack; thromboembolism; Prevention and control
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Low dose
  Interventions: Drug: YM150
- 2 (Experimental): Middle dose
  Interventions: Drug: YM150
- 3 (Experimental): High dose
  Interventions: Drug: YM150
- 4 (Active Comparator)
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: YM150 — Oral
  Arms: 1; 2; 3
Drug: warfarin — Oral
  Arms: 4

SUMMARY:
To evaluate the safety and tolerability of YM150 in subjects with non-valvular atrial fibrillation (NVAF)and to obtain information on pharmacokinetics and pharmacodynamics (anti-thrombotic potential) in the target population

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for the study if all of the following apply:

* Subject has paroxysmal permanent or persistent NVAF
* Subject has INR of 2.0 or below and an aPTT ≤ 1.5 times the upper limit of normal at the baseline visit.
* Legal minimum age requirement (country-specific).
* Written informed consent has been obtained.

Exclusion Criteria:

* History of heart valve disorders
* History of rheumatic fever.
* History of stroke and/or systemic embolism (including TIA).
* History of Acute Coronary Syndrome (ACS).
* Indication for warfarin other than NVAF.
* Known hemorrhagic disorder and/or coagulation disorder.
* Active bleeding or any condition associated with increased risk of bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
All clinically relevant bleeds during the treatment period rated as "major" or "clinically relevant non-major(CRNM)" | 16 Weeks

SECONDARY OUTCOMES:
Incidence of symptomatic stroke | 16 Weeks
Incidence of transient ischemic attack (TIA) | 16 Weeks
Incidence of systemic thromboembolic event | 16 Weeks
Incidence of the bleeding rates | 16 Weeks
Other safety assessments | 16 Weeks
PK, PD variables | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (18):
- Launceston, Australia
- Hong Kong (2):
  - Pok Fu Lam
  - Shatin
- Japan (6):
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Shikoku
  - Tōhoku
- Kuala Lumpur, Malaysia
- Hastings, New Zealand
- Singapore, Singapore
- Bloemfontein, South Africa
- Seoul, South Korea
- Taipei, Taiwan
- Thailand (3):
  - Bangkok
  - Chiang Mai
  - Nakhon Ratchasima